CLINICAL TRIAL: NCT06808386
Title: Comparison of the Effects of Different Training Frequencies on the Rehabilitation of Individuals with Patellofemoral Pain: a Randomized Clinical Trial
Brief Title: Effects of Training Frequency on Patellofemoral Pain Rehabilitation.
Acronym: ETFRPPRRCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Paulo Roberto Garcia Lucareli, Head of Human Movement Analysis Laboratory, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 84694624.0.0000.5511
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Anterior Knee Pain
Keywords: Patellofemoral Pain; Exercise Therapy; Dose-Response; Musculoskeletal Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strengthening 2 times per week (Experimental): This group will consist of participants with patellofemoral pain and will receive treatment twice a week.
  Interventions: Other: Strengthening 2 times per week
- Strengthening 3 times per week (Other): This group will consist of participants with patellofemoral pain and will receive treatment twice a week.
  Interventions: Other: Strengthening 3 times per week

INTERVENTIONS:
Other: Strengthening 2 times per week — This group will consist of participants with patellofemoral pain and will receive treatment twice a week.
  Arms: Strengthening 2 times per week
Other: Strengthening 3 times per week — This group will consist of participants with patellofemoral pain and will receive treatment thrice a week.
  Arms: Strengthening 3 times per week

SUMMARY:
This clinical trial aims to determine the optimal frequency of exercise therapy for improving pain, function, and quality of life in participants with patellofemoral pain. The main questions it aims to answer are:

Does exercising twice a week provide the same benefits as exercising three times a week for individuals with patellofemoral pain? What are the optimal dosage, volume, and weekly exercise frequency for treating patellofemoral pain?

The investigators will compare two groups of participants: one group of participants receiving exercise therapy twice a week and another group receiving exercise therapy three times a week. Both groups will follow the same exercise protocol targeting the muscles of the hip and knee joints.

Participants:

84 volunteers (both male and female) with patellofemoral pain Physically active individuals aged between 18 and 40 years

Interventions:

Participants will be randomly assigned to one of two groups Both groups will perform the same exercises for hip and knee muscle strengthening Group A will exercise three times per week Group B will exercise two times per week The intervention will last for six consecutive weeks

Assessments: Participants will be evaluated at the following time points:

Before the intervention After the 4th and 6th week of intervention 6 months and 1 year after the end of the intervention

The primary Outcome Measure will be pain intensity.

Secondary Outcome Measure:

Anterior knee pain during daily activities Kinesiophobia Pain-related self-efficacy Chronic pain-related self-efficacy Catastrophizing Muscle strength 3D Movement analysis

Data Analysis:

The investigators will use an intention-to-treat analysis, which means that all participants will be included in the study, regardless of whether they completed the treatment as planned.

Appropriate statistical tests will be used to compare differences within and between the two groups, considering the time points and group factors.

A 5% significance level will be adopted, which means there is a 5% chance that the results are due to random variation rather than the treatment effect.

DETAILED DESCRIPTION:
This clinical trial aims to investigate the optimal frequency of exercise therapy for individuals with patellofemoral pain. Current evidence supports exercise therapy as the first line of treatment for pain relief, improved function, and enhanced quality of life in individuals with patellofemoral pain. However, the most recent consensus on patellofemoral pain highlighted a gap in the ideal dosage, volume, and weekly exercise frequency for treating these individuals.

To address this gap, this study will compare two groups of individuals with patellofemoral pain who will undergo the same exercise program targeting the muscles of the hip and knee joints but with different frequencies. One group will perform the exercises twice weekly, while the other will do so thrice.

This randomized, controlled, double-blind clinical trial will recruit 84 physically active participants of both sexes, aged 18 to 40 years, who experience patellofemoral pain. Participants will be randomly and secretly allocated to one of two groups. Group A will perform the exercise protocol three times per week, and Group B will perform the same protocol twice weekly.

The intervention will last for six consecutive weeks. Participants will be evaluated at multiple time points: before the intervention, after the 4th and 6th week of intervention, and at 6 months and 1 year post-intervention. The evaluations will include pain intensity as a primary outcome, anterior knee pain during daily activities, kinesiophobia, pain-related self-efficacy, chronic pain-related self-efficacy, catastrophizing, muscle strength and 3d movement analysis as a secondary analysis.

The data analysis will follow the intention-to-treat principle, meaning all participants will be included in the analysis regardless of whether they completed the treatment as planned. Normality tests will be conducted to verify data distribution, and appropriate statistical tests will be used to compare differences within and between the two groups, considering time and group factors. A 5% level of significance will be adopted for statistical comparisons.

ELIGIBILITY:
Inclusion Criteria: This study will include physically active individuals of both sexes, aged between 18 and 40 years, who have been experiencing patellofemoral pain and anterior knee pain for at least three months. Participants must have a score of at least three points on the Visual Analog Scale during any of the following activities: running, squatting, sitting for long periods with the knee bent, and climbing or descending stairs. Selection will be based on responses provided in the International Physical Activity Questionnaire.

Exclusion Criteria: Exclusion criteria include the following: a history of lower limb or spine surgery, patellar dislocation, anterior knee pain resulting from trauma, coexisting conditions in the knee joint such as meniscal and/or ligament injuries, lateral and/or posterior knee pain, cardiovascular issues or locomotion disorders that could impact the assessment, pregnancy, and a limb length discrepancy greater than 1 cm.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Evaluations will occur at five time frames: 24 hours before the first treatment session, after the 4th and 6th weeks of treatment, and 6 months and 1 year after the last session.
  Visual Analog Pain Scale: This scale aims to quantify the intensity of pain experienced by the patient. The scale consists of 11 points, with a score classification from 0 to 10. A score of 0 represents "no pain at all", and 10 means "the worst pain possible". Patients will be asked to rate their anterior knee pain intensity levels based on the past fifteen days. The minimum clinically important difference for improvement will be a decrease of 1 point on the scale.

SECONDARY OUTCOMES:
Anterior Knee Pain Scale | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment, and 6 months and 1 year after the last session.
  This is a specific questionnaire for anterior knee pain, consisting of 13 items categorised into different knee function levels. Each item is answered, and the total result is added to a global index with a maximum score of 100 points, representing "no deficit," and a minimum score of zero, representing "the greatest possible deficit". The minimum clinically significant difference for improvement will be a reduction of 2 points on the scale.
Tampa Scale for Kinesiophobia | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment, and 6 months and 1 year after the last session.
  This psychometric questionnaire quantifies the fear associated with pain. It consists of 17 questions, each scored on a four-point Likert scale. The total score ranges from 17 to 68 points, with values above 37 points indicating a higher fear associated with movement.
Pain Self-Efficacy Questionnaire | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment, and 6 months and 1 year after the last session.
  This psychometric questionnaire quantifies the patient's confidence in performing activities despite pain. It consists of ten questions, each scored on a six-point Likert scale. The total score ranges from 10 to 60 points, with higher values indicating greater patient confidence regardless of pain.
Chronic Pain Self-Efficacy Scale | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment, and 6 months and 1 year after the last session.
  This psychometric scale consists of 22 items that measure the confidence of patients with chronic pain in performing specific tasks in different domains: pain control, physical function, and symptom control. Each item is scored on a Likert scale ranging from ten to 100 points, with higher values indicating greater patient confidence regardless of pain.
Pain Catastrophizing Scale | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment, and 6 months and 1 year after the last session.
  This questionnaire consists of 13 statements that contain various thoughts and feelings a person may have when experiencing pain. The items are divided into rumination, magnification, and helplessness, each scoring on a 5-point scale. Participants are asked to rate how often they experience these feelings, from 0 (not at all) to 4 (always). The total score ranges from 0 to 52 points, with higher scores indicating greater pain catastrophizing.
Global Perceived Effect Scale | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment, and 6 months and 1 year after the last session.
  The perception of the global effect of the treatment by the research participant will be assessed using the Global Perceived Effect Scale. The Global Perceived Effect Scale is a direct scale, validated for Brazilian Portuguese, with good psychometric properties, which aims to assess self-perception of the intervention performed. Participants will be asked: "Compared to the beginning of the treatment, how would you describe your knee(s) today?" Participants will then mark their response on an 11-point scale, ranging from -5 (worse than before treatment), 0 (neutral), to +5 (better than before treatment). The minimum clinically important difference for improvement will be 2.5 points on the scale (Freitas et al., 2019; Bobos et al., 2020).
Maximum isometric muscle strength | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment.
  Maximum isometric muscle strength measure maximum isometric muscle strength using a manual dynamometer.
Three-dimensional movement analysis | 24 hours before the first treatment session, after the 4th and 6th weeks of treatment
  Three-DimensionalMovement Analysis is a comprehensive technique used to evaluate the movement and forces involved in body motions.
  Kinematic analysis focuses on the motion of body segments and joints in three dimensions, capturing data on their positions, velocities, and accelerations.
  Kinetic analysis examines the forces that cause these movements, such as muscle forces, ground reaction forces, and joint moments.
  By combining both kinematic and kinetic data, this analysis provides a detailed understanding of the biomechanics of human motion.

CONTACTS AND LOCATIONS:
Overall Officials: PAULO RG LUCARELI, PhD, Study Chair — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No